CLINICAL TRIAL: NCT04194476
Title: Performance Study of Nova StatStrip® Blood Glucose Monitoring Test System on Neonatal Capillary Blood
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The protocol needs to be further developed.
Sponsor: Nova Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NB15-CHI-SSG-NEO
Record Dates: First submitted 2019-12-06; First posted 2019-12-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Healthy and Unhealthy Neonates
Keywords: neonates; glucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- 120 neonates less than 28 days old (Experimental): Each neonate will be tested for blood glucose level twice on the same heel stick site using two glucose meters. additional 200-300 ul blood will be collected and centrifuged. Plasma will be tested blood glucose in the lab analyzer in the clinical laboratory.
  Interventions: Diagnostic Test: StatStrip blood glucose meter and strips

INTERVENTIONS:
Diagnostic Test: StatStrip blood glucose meter and strips — We'll use a drop of heel-stick blood to test blood glucose on the glucose meter. About 200-300 ul of blood from the same stick site will be collected, centrifuged to get plasma for testing of glucose level in a laboratory biochemistry analyzer.

SUMMARY:
This study is to determine the validity of Nova StatStrip® blood glucose monitoring test system including the Nova StatStrip® glucose hospital meter and test strips in measuring Chinese neonatal capillary blood glucose levels by evaluating how the results compare to those obtained from laboratory hexokinase method. The study results will be the basis for the regulatory submission and registration of the Nova StatStrip® glucose hospital meter and test strips in testing the neonatal capillary whole blood specimens to the China Food and Drug Administration (CFDA).

Good clinical practice indicates that the performance of a point-of-care glucose monitoring test system be validated before clinical use. It is therefore important to perform a method comparison study to determine how the results obtained from a type of glucose monitoring test system compare to those from a laboratory hexokinase method.

ELIGIBILITY:
Inclusion Criteria:

* Subject is within 28 days after birth.
* The legal representative of the Subject agrees to sign two copies of the Informed Consent Form.
* The Subject's capillary whole blood needs to be drawn via heel stick for routine clinical laboratory testing according to the prescription.
* The legal representative of the Subject agrees that the Subject provides 300 µL capillary whole blood for glucose and haematocrit testing in addition to routine clinical laboratory testing.

Exclusion Criteria:

* Subject/legal representative is currently working for, has previously worked for, or has an immediate family member working for a company manufacturing and/or marketing blood glucose monitoring products;
* Subject has already participated in this study.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
blood glucose level measured by StatStrip blood glucose meter | 6 months
plasma glucose level measured by a laboratory biochemistry analyzer | 6 months

SECONDARY OUTCOMES:
hematocrit of the heel-stick blood | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China